CLINICAL TRIAL: NCT01510236
Title: A Randomized Controlled Study of the Clinical Efficacy and Cost-effectiveness of a Self-help Program Via Internet on Psychosocial Function Among Adolescents With Cancer
Brief Title: Self-help Program Via Internet for Adolescents With Cancer
Acronym: U-CARE:TeenCan
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: a feasibility study showed low recruitment and adherence
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Louise-von Essen, Professor, Programme Director for U-CARE, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: U-CARE: TeenCan
Record Dates: First submitted 2012-01-04; First posted 2012-01-16 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Cancer; Depression; Anxiety
Keywords: Adolescence; Cancer; Depression; Anxiety; Self-help via internet
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders

ARMS (2):
- Early self-help program (Experimental): The early self-help program starts directly after randomization i.e. 4 weeks after diagnosis.
  Interventions: Behavioral: Self-help program
- Later self-help program (Experimental): The later self-help program starts sixty-two weeks after diagnosis.
  Interventions: Behavioral: Self-help program

INTERVENTIONS:
Behavioral: Self-help program — The program is available via an internet platform (www.carebase.se) and consists of two steps: interactive support (Step 1) and cognitive behavioral therapy (CBT) delivered via internet (2). Step 1 provides information about the cancer experience and psychoeducation about frequent reactions and distress and how to manage this. The information and education is provided via texts, audio files, and video-interviews with persons who have survived cancer during adolescence. Step 1 also capitalizes on interaction between participants via chat and forum. There is also a possibility to ask questions to an expert via the website. Twenty-eight weeks after start of Step 1 participants are offered access to Step 2 which lasts ten weeks and consists of a self-help CBT material consisting of modules and weekly contact with a psychologist. Each module is focused on one problem area, e.g. worry or depressive symptoms. Step 1 is available during Step 2. The whole program lasts for 34 weeks.

SUMMARY:
The overall aim is to evaluate the clinical efficacy and cost-effectiveness of a self-help program via internet aiming at preventing development and maintenance of cancer-related emotional distress among adolescents with cancer.

DETAILED DESCRIPTION:
A significant number of adolescents reports less anxiety and depression and a better quality of life than a healthy reference group from eighteen months up to four years after diagnosis. However, a significant minority of adolescents struck by cancer reports a clinically relevant level of emotional distress from shortly after diagnosis up to four years after diagnosis. The provided self-help program is designed to promote psychological health.

150 adolescents recently diagnosed with cancer will be randomized to either of two conditions: (1) Early program and (2) Later program. In both conditions an internet-based self-help program is provided. Adolescents randomized to Early program start the program directly after randomization i.e. 4 weeks after diagnosis whereas adolescents randomized to Later program start the program sixty-two weeks after diagnosis. The larger part of data are collected at seven assessments, Observations 1-7. Observation 1 takes place 4 weeks after diagnosis (DI); Observation 2: 28 weeks after DI; Observation 3: 38 weeks after DI; Observation 4: 62 weeks after DI; Observation 5: 86 weeks after DI; Observation 6: 96 weeks after DI and Observation 7: 120 weeks after DI. The main research question is to investigate whether the program is superior to standard care in preventing development and maintenance of anxiety and depression at 38 weeks after diagnosis among adolescents with cancer.

ELIGIBILITY:
Inclusion criteria:

* Adolescents aged from 13 to 19
* Recent cancer diagnosis

Exclusion criteria:

* No access to computer or internet
* Difficulties reading or understanding Swedish

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Observation 3 (38 weeks after DI)

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist - Civilian Version (PCL-C) | Observation (OBS) 1: 4 weeks after diagnosis (DI); OBS 2: 28; OBS 3: 38; OBS 4: 62; OBS 5: 86; OBS 6: 96 and OBS 7: 120 weeks after DI.
UCLA Loneliness Scale | Observation (OBS) 1: 4 weeks after diagnosis (DI); OBS 2: 28; OBS 3: 38; OBS 4: 62; OBS 5: 86; OBS 6: 96 and OBS 7: 120 weeks after DI.
Rosenberg Self-Esteem Scale (RSE) | Observation (OBS) 1: 4 weeks after diagnosis (DI); OBS 2: 28; OBS 3: 38; OBS 4: 62; OBS 5: 86; OBS 6: 96 and OBS 7: 120 weeks after DI.
Satisfaction With Life Scale (SWLS) | Observation (OBS) 1: 4 weeks after diagnosis (DI); OBS 2: 28; OBS 3: 38; OBS 4: 62; OBS 5: 86; OBS 6: 96 and OBS 7: 120 weeks after DI.
Mental Health Continuum - Short form (MHC-SF) | Observation (OBS) 1: 4 weeks after diagnosis (DI); OBS 2: 28; OBS 3: 38; OBS 4: 62; OBS 5: 86; OBS 6: 96 and OBS 7: 120 weeks after DI.
EQ-5D | Observation (OBS) 1: 4 weeks after diagnosis (DI); OBS 2: 28; OBS 3: 38; OBS 4: 62; OBS 5: 86; OBS 6: 96 and OBS 7: 120 weeks after DI and 6, 8, 12, 16, 20, 24, 29, 33, 37, 38, 64, 66, 70, 74, 78, 82, 87, 91, and 95 weeks after DI.
  Quality of life for parents and adolescents
Posttraumatic Growth Inventory - Short form (PTGI-SF) | Observation (OBS) 3: 38 weeks after diagnosis (DI); OBS 4: 62; OBS 6: 96 and OBS 7: 120 weeks after DI.
Health-related costs questionnaire | Observation (OBS) 2: 28 weeks after diagnosis (DI); OBS 3: 38; OBS 4: 62; OBS 5: 86; OBS 6: 96 and OBS 7: 120 weeks after DI and 8, 16, 66, and 74 weeks after DI.
  Measurement of health-related costs for parents and adolescents such as sick-leave, transports, health-care visits, consumption of medicines etc.
Time spent on self-help program | Observation (OBS) 1: 4 weeks after diagnosis (DI); OBS 2: 28; OBS 3: 38; OBS 4: 62; OBS 5: 86; OBS 6: 96 and OBS 7: 120 weeks after DI.
  Measurement of hours spent on program (time cost)

CONTACTS AND LOCATIONS:
Overall Officials: Louise von Essen, PhD, Principal Investigator — Uppsala University
Locations (6):
- Sweden (6):
  - Drottning Silvias Barn- och Ungdomssjukhus, Gothenburg
  - Universitetssjukhuset, Linköping
  - Barn- och Ungdomssjukhuset, Lund
  - Astrid Lindgrens Barnsjukhus, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Barnsjukhuset, Uppsala

REFERENCES:
- See also: U-CARE — http://www.u-care.uu.se/?languageId=1